CLINICAL TRIAL: NCT04128826
Title: Effect of Triceps Range of Motion Exercise on Shooting Accuracy Among Recreational Basket Ball Players
Brief Title: Triceps Range of Motion Exercise on Shooting Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UMFD3026
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Recreational Basket Ball Players
Keywords: Partial Range of Motion; Full Range of Motion
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent individual outcome assessor will not know participants belongs to which group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Partial Range of Motion (PROM) (Experimental)
  Interventions: Other: Resistance Training
- Full Range of Motion (FROM) (Experimental)
  Interventions: Other: Resistance Training
- Control (CON) (No Intervention)

INTERVENTIONS:
Other: Resistance Training — Using the cable machine, shoulders will be flexed to 180° for both (PROM & FROM) groups throughout the training; FROM would train with full elbow extension (complete elbow flexion to extension) whereas PROM will train with partial elbow extension from 60° to 110°. A total of 8 sessions, 2 sessions/week for 4 weeks will be carried out by both groups. CON group will not participate in training protocol.
  Arms: Full Range of Motion (FROM); Partial Range of Motion (PROM)

SUMMARY:
Theories support that nearly all the movements performed by athletes- from rebounding to steal the basketball, to riding a bicycle occur within a small range of motion and training in partial range can improve the isometric strength within the range of motion which it is trained and also increase the full range of motion (FROM) strength as well. The best training method to improve the shooting accuracy among basketball players remains unclear, despite the numerous training methods being available. The aim of this study is to compare the effect of tricpes full range of motion vs triceps partial range of motion training on shooting accuracy among recreational basket ball players. The previous research has mostly focused on measuring the isokinetic strength at different speed in relation to shooting accuracy and there is limited research which has explored the triceps strength using partial range exercise.

DETAILED DESCRIPTION:
Optimally designed exercise protocols for weight training are are based on scientiﬁc principles which manipulate essential training variables, including the order of the exercise, frequency, volume, intensity, rest intervals between sets, and others. The distance covered by the repetition that is carried out within a restricted part of a repetition is defined as a partial repetition (PR). The starting range of motion or range which is close to full range of the repetition are most commonly focused in most cases of sports training's. It is because of the muscle length-tension relationship, activation of the muscle and total mass of muscle, the muscle strength which is produced by full range of the movement of any particular joint will vary. In resistance training, the training range is most beneficial and effective if the repetition is stopped right before the full contraction is achieved, as this stopping prevents the load being always applied to the working muscle. For some of the exercises, the risk of a muscle tear is increased by the point of total contraction on the negative movement because muscle fibers are stretched way beyond the control point. Partial range of motion (PROM) is a mode of training which is not a recent finding and has projected some beneficial effects and efﬁciency in improving the outcomes in addition of improving the isometric strength. When the shoulder is elevated beyond 90°, the medial head of the triceps is activated the most. During basketball shooting, the medial head of triceps is important as the shoulder elevation is more than 90° when performing a jump shooting. According to this analysis of muscle force and activation of each head of triceps in relation to motion of shoulder elevation and elbow angle, it shows that medial head is most activated at 180° of shoulder elevation and between 60° to 110° of elbow extension. Thus, it can be suggested that when performing a jump shooting with shoulder elevation more than 90°, the medial head of triceps helps in forceful extension of arm to throw the basketball. PROM resistance training is proven to have positive effects in strength gain in various ranges and isokinetic strength of triceps that are correlated with shooting accuracy. This study will investigate the effectiveness of FROM and PROM training in improving shooting accuracy as there is dearth in current literature on triceps isotonic strength of different range of motion on shooting accuracy. This will be a single blinded randomized control trial study and a total of male 30 participants would be recruited using purposive sampling method. Participants will be assigned into three groups; FROM, PROM and control group (CON). Using the cable machine, shoulders will be flexed to 180° for both groups throughout the training; FROM will train with full elbow extension (complete elbow flexion to extension) whereas PROM would train with partial elbow extension from 60° to 110°. Both groups will perform at 67% of 1 repetition maximum with 10 repetition in one set, and a total of 4 sets will be carried out by each group. A rest period of 2 minutes will be permitted between sets. A total of 8 sessions, 2 sessions/week (muscle soreness is reduced greatly after 72 hours of rest after exercise will be carried out by both groups. CON group will not participate in training protocol. All the participants will be tested as baseline and at the end of four weeks training using three point shooting (S3P). The shooting accuracy will be measured using S3P method. The subjects will be required to perform 3 sets of the test to get an average score. There will be 5 positions marked on the basketball court, each point at a distance of 6.25m away from the hoop. The first point will be set at the right wing of the court, which is at 0° to the hoop, the second point will be set 45° away from the first point, and also 6.25 m from the hoop, third point at 90°, facing the board and the hoop, also marked 6.25 m away from the hoop. The 4th and 5th point will be similar to 1st and 2nd point, just that the points will be marked to the left side of the court. Each player will shot for 10 points in one set, 2 points from each point.

ELIGIBILITY:
Inclusion Criteria:

* Male Recreational Basket Ball Players
* Age 18 to 25 years
* Height 1.7 to 1.8 meters

Exclusion Criteria:

* Female Gender
* Professional Basket Ball Payers
* Presence of Musculo-skeletal Injury in past 6 months
* Performance enhancing Drugs
* Any influence of any Medication that can affect Balance and Co-ordination

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
three point shooting (S3P) | At baseline (before intervention begun) and 1 day post 4 weeks of training
  The shooting accuracy will be measured via 3 attempts of S3P method. The subjects will be required to perform 3 sets of the test to get an average score. 5 positions will be marked on the basketball court, each point 6.25m away from the hoop. The first point would be set at the right wing of the court, which is at 0° to the hoop, the second point will be set 45° away from the first point, and also 6.25 m from the hoop, third point at 90°, facing the board and the hoop, also marked 6.25 m away from the hoop. The 4th and 5th point will be similar to 1st and 2nd point, just that the points would be marked the left side of the court. Each player will shot for 10 points in one set, 2 points from each point.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

REFERENCES:
- [Background] Pinto RS, Gomes N, Radaelli R, Botton CE, Brown LE, Bottaro M. Effect of range of motion on muscle strength and thickness. J Strength Cond Res. 2012 Aug;26(8):2140-5. doi: 10.1519/JSC.0b013e31823a3b15. PMID 22027847
- [Background] Richardson, K. (2013). Partial Reps vs Full Range Of Motion- What Works Best?. Naturally Intense Diet & Fitness Blog. Retrieved 10 October 2018. https://naturallyintense.net/blog/exercise/weight-training/partial-reps-vs-full-range-of-motion-what-works-best/
- [Background] Locke B (2005). Effective Full Range of Motion. Bodybuilding.com. Retrieved 10 October 2018. https://www.bodybuilding.com/fun/teen-locke3.htm
- [Background] Newmire DE, Willoughby DS. Partial Compared with Full Range of Motion Resistance Training for Muscle Hypertrophy: A Brief Review and an Identification of Potential Mechanisms. J Strength Cond Res. 2018 Sep;32(9):2652-2664. doi: 10.1519/JSC.0000000000002723. PMID 29985227
- [Background] Massey CD, Vincent J, Maneval M, Moore M, Johnson JT. An analysis of full range of motion vs. partial range of motion training in the development of strength in untrained men. J Strength Cond Res. 2004 Aug;18(3):518-21. doi: 10.1519/13263.1. PMID 15320644
- [Background] Kholinne E, Zulkarnain RF, Sun YC, Lim S, Chun JM, Jeon IH. The different role of each head of the triceps brachii muscle in elbow extension. Acta Orthop Traumatol Turc. 2018 May;52(3):201-205. doi: 10.1016/j.aott.2018.02.005. Epub 2018 Mar 2. PMID 29503079
- [Background] Baechle, T., R. Earle, And D. Wathen (2016) . Resistance training. In: Essentials of Strength Training and Conditioning.T.R.Baechle and R.W. Earle, eds. Champaign, IL: Human Kinetics, 2000. pp. 395-425.
- [Background] Baroni BM, Pompermayer MG, Cini A, Peruzzolo AS, Radaelli R, Brusco CM, Pinto RS. Full Range of Motion Induces Greater Muscle Damage Than Partial Range of Motion in Elbow Flexion Exercise With Free Weights. J Strength Cond Res. 2017 Aug;31(8):2223-2230. doi: 10.1519/JSC.0000000000001562. PMID 27398917
- [Derived] Mir IA, Mohd Jamali MNZ, Humayra S, Chong KW, Amalnerkar T, Sirajudeen MS. Partial versus full range of motion triceps strength training on shooting accuracy among recreational basketball players: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Mar 6;17(1):41. doi: 10.1186/s13102-025-01060-2. PMID 40051008